CLINICAL TRIAL: NCT06125457
Title: Epidemiology of IgA Selective Deficiency - Clinical Manifestations and Risk of Transmission: A Retrospective Cohort Study in Strasbourg University Hospital
Brief Title: Epidemiology of IgA Selective Deficiency - Clinical Manifestations and Risk of Transmission
Acronym: EpIgA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8587
Record Dates: First submitted 2022-09-01; First posted 2023-11-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: COVID-19; IgA deficiency; Antibiotic therapy; Immunosuppressive treatments; Autoimmune manifestations; Neoplasia
MeSH Terms: conditions — COVID-19; IgA Deficiency; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of patients with a selective IgA deficiency currently consists of symptomatic treatment with treatment of infections by occasional or prolonged antibiotic therapy, immunosuppressive treatments for autoimmune pathologies, symptomatic treatment of allergic manifestations.

IVIG supplements are sometimes proposed in the event of recurrent infections and the demonstration of deficiencies in IgG subclasses (IgG1, 2, 3) often not sought for diagnosis The factors associated with the severity of clinical manifestations are not well identified and patients with IgA deficiency must be monitored over the long term because of the risk of the appearance of autoimmune manifestations and neoplasia. The identification of such factors could lead to the proposal of close monitoring for these patients.

IgA deficiency, which is frequent, has not been identified as a risk factor for severe COVID-19 infection, probably due to a lack of studies with sufficient recruitment. The therapeutic attitude concerning patients with an IgA deficiency in the event of COVID-19 infection is therefore not consensual.

There is currently no action to be taken regarding the risk of transmission of IgA deficiency.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject treated at the HUS, with a primary selective IgA deficiency, considered as definitive (IgA concentration < 0.07g/L or total absence of IgA on immunofixation) or as probable (IgA concentration lower than two standard leads to standard for age) with no other humoral immunodeficiency and no other cause of decreased gammaglobulins 01/01/2005 to 01/31/2022.
* Subject having not expressed, after being informed, their opposition to the reuse of their data for the purposes of this research.

Exclusion criteria:

. Subject who expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) with a primary selective IgA deficiency treated at the HUS from 01/01/2005 to 01/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-09 (Actual); Primary Completion 2023-12-09 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive test result for covid-19 | 1 hour after hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Immunologie Clinique - Médecine Interne - CHU de Strasbourg - France, Strasbourg, France